CLINICAL TRIAL: NCT03339908
Title: Regional Non-comparative Prospective Study of the Impact of Gamma Knife Radiosurgery on Tremor in Multiple Sclerosis
Acronym: GK-SEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-22; 2016-A01071-50 (Registry Identifier: ID RCB)
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with Multiple Sclerosis (Experimental): Patients will benefit from unilateral thalamotomy by Gamma Knife radiosurgery
  Interventions: Device: Thalamotomy by gamma Knife radiosurgery

INTERVENTIONS:
Device: Thalamotomy by gamma Knife radiosurgery — The surgical procedure consists of a very partial radiation of the brain with stereotaxic precision

SUMMARY:
Multiple sclerosis, chronic inflammatory disease of the central nervous system, affects approximately 100,000 peoples in France. It is the leading cause of disability in young adults. Tremor is a common symptom (25-58% of patients depending on the series) and can be particularly disabling. The drug treatments against tremor are ineffective or insufficient. Deep brain stimulation of the Vim (Small nucleus within thalamus) and stereotactic radiofrequency thalamotomy have shown their efficacy in this indication. However, in some cases these invasive procedures are impossible because of operational risk. Gamma knife thalamotomy can be an alternative choice. This procedure, less invasive, mainly because of the absence of craniotomy is used by several teams of international reputation for over fifteen years, with good to excellent results in essential tremor. The team of Marseille, which has an experience of 22 years in Gamma Knife radiosurgery has treated 250 patients with severe tremor (essential tremor or Parkinson's disease) by a unilateral thalamotomy with an improvement of 70% of functional scores.

In the literature, no formal studies of the effect of Gamma Knife in Multiple Sclerosis (MS) tremor is reported. There are only a few cases without specific evaluation of the efficacy in this disease. Hence the importance of studying in detail the effects of this technique, which allows a precise and limited lesion volume. Using an isocenter of 4mm and a dose of 130 Gy radiation lesion obtained is limited to a volume of 200 to 500 mm3.

The aim of this study is to assess through a minimally invasive technique with a circumscribed and reproducible lesion volume, the effect of thalamotomy on the particular tremor in multiple sclerosis with a prospective evaluation of its effects.

Patients with MS with a disabling tremor will be included in the study. They will be assessed with neurological examination, quality of life scales, neuropsychological assessment, functional scores and cerebral MRI.

This study will demonstrate the feasibility and effectiveness of Gamma Knife thalamotomy in MS patients with severe tremor.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 70 years old.
* Patient with a diagnosis of MS certainty according to the criteria of Mac Donald (2010)
* Patient with progressive form of MS: remitting, secondarily progressive, primary progressive
* Patient with an Expanded Disability Status Scale score (EDSS) between 3 and 8.
* Patient with clinical stability for more than 6 months (EDSS stable over 1 year)
* Lack of progressive onset (and corticosteroid therapy) for at least 3 months
* Patient with normal palliation or mild impairment
* Patient having a muscle test at 4 or 5 on the upper limb to be treated
* Patient requiring Gamma-Knife radiosurgery due to severity of tremor and functional impairment
* Patient who understood and signed the informed consent form

Exclusion Criteria:

* Stewart Holmes positive maneuver (upper limb to be treated)
* Patient with a muscle test less than 4 on the hand to be treated
* Patient with moderate palliation or severe disease
* Patient with a contraindication to perform a cerebral MRI (pacemaker, intracerebral metallic object etc.)
* Patient with an indication for radiosurgical treatment
* Pregnant or lactating women.
* Participation in another therapeutic trial or exclusion period from a previous clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Scale evaluation Tremor and Coordination Scale (TACS) | 12 months
  Describe the effectiveness of the Gamma Knife radiosurgical treatment. Assess the impact of tremor and impaired coordination on daily activities. The TACS was developed as a single question, scored ordinally from 0 to 5, as follows: 0 (normal), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe), or 5 (total disability). This scoring system makes it similar to the Performance Scales
Scale evaluation Tremor and Coordination Scale (TACS) | 24 months
  Describe the effectiveness of the Gamma Knife radiosurgical treatment. Assess the impact of tremor and impaired coordination on daily activities. The TACS was developed as a single question, scored ordinally from 0 to 5, as follows: 0 (normal), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe), or 5 (total disability). This scoring system makes it similar to the Performance Scales

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marie REGIS, PU-PH, Principal Investigator — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided